CLINICAL TRIAL: NCT07150923
Title: Comparing Two Multicomponent Strategies To Promote Supraglottic Airway Implementation During Neonatal Resuscitation
Brief Title: Supraglottic Airway for Resuscitation Trial
Acronym: SUGAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-022884; 33954 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Resuscitation; Delivery Room Resuscitation; Positive Pressure Ventilation; Infant, Newborn; Supraglottic Airway; Laryngeal Mask Airways; Implementation Research
Keywords: Neonatal Resuscitation; Delivery Room Resuscitation; Positive pressure ventilation; Supraglottic Airway; Laryngeal Mask Airways; Implementation Research; Infant, Newborn

STUDY DESIGN:
Intervention Model Description: Hybrid type 3 effectiveness-implementation parallel cluster randomized superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard of Care ("Enhanced") (Active Comparator)
  Interventions: Other: Enhanced Standard of Care ("Enhanced")
- Enhanced Standard of Care Plus Facilitation ("Enhanced-Plus") (Active Comparator)
  Interventions: Other: Enhanced Standard of Care ("Enhanced-Plus")

INTERVENTIONS:
Other: Enhanced Standard of Care ("Enhanced") — Enhanced Standard of Care ("Enhanced") will include: Educational Materials and Outreach, Local Champions, Train the Trainer, Local Simulation Training, and SA Starter Packs.
  Arms: Enhanced Standard of Care ("Enhanced")
Other: Enhanced Standard of Care ("Enhanced-Plus") — Enhanced Standard of Care ("Enhanced-Plus") will include: Educational Materials and Outreach, Local Champions, Train the Trainer, Local Simulation Training, SA Starter Packs, and three additional intensive external facilitation components.
  Arms: Enhanced Standard of Care Plus Facilitation ("Enhanced-Plus")

SUMMARY:
This is a hybrid type 3 effectiveness-implementation parallel cluster randomized superiority trial designed to compare two strategies to promote early supraglottic airway (SA) rescue during neonatal resuscitation, with a focus on implementation outcomes.

DETAILED DESCRIPTION:
Each year, approximately 3.8 million infants are born in the United States, and up to 10% require resuscitation to establish breathing at birth. Positive pressure ventilation (PPV) is the most important intervention during neonatal resuscitation and is most often delivered via facemask. However, facemask ventilation can be technically challenging, and difficulties with mask seal, airway positioning, and obstruction frequently lead to ventilation failure. Such delays prolong life-threatening asphyxia and increase the risk of morbidity and mortality.

The supraglottic airway (SA) is an FDA-approved, widely available, and evidence-based alternative airway device for delivering PPV. It is safe, easy to use, and recommended in international neonatal resuscitation guidelines as an option when facemask ventilation is ineffective or endotracheal intubation is unsuccessful or not feasible. Despite strong supporting evidence, uptake of SA use in neonatal resuscitation remains low. A recent national survey of more than 5,000 Neonatal Resuscitation Program (NRP) providers found that only 12% had ever used an SA. Reported barriers to adoption included limited clinical experience, insufficient training opportunities, preference for alternative approaches, lack of availability of SA devices in the delivery room, and limited awareness of supporting evidence.

The Supraglottic Airway for Resuscitation (SUGAR) Trial is designed to address the critical evidence-to-practice gap by evaluating strategies to increase the use of supraglottic airways (SA) during neonatal resuscitation. This trial will assess the comparative effectiveness of two implementation strategies while examining the contextual factors that influence their success, with the goal of identifying barriers and facilitators to sustainable SA adoption across diverse clinical settings. By testing approaches to integrate SA use into routine neonatal resuscitation, the study aims to improve both implementation and clinical outcomes, ultimately reducing the risk of prolonged asphyxia and enhancing survival and health for newborns in the delivery room.

ELIGIBILITY:
Population 1: Hospital Staff

Population 1a: Clinical providers and administrators who complete study questionnaires

Clinical provider 1a inclusion criteria:

* Employed full-time by the hospital, affiliated practice, or affiliated university in a role that involves newborn resuscitation
* Fluent in English

Administrator 1a inclusion criteria

* Oversee the care of newborns on a local level (e.g. nurse manager) or a hospital level (e.g. Chief Quality and Safety Officer)
* Fluent in English

Clinical provider and administrator exclusion 1a criteria: No exclusion criteria

Population 1b: Clinical providers who participate in qualitative interviews

Clinical provider 1b inclusion criteria:

* Employed full-time by the hospital, affiliated practice, or affiliated university in a role that involves newborn resuscitation
* Fluent in English

Clinical provider 1b exclusion criteria: No exclusion criteria

Population 2: Patients who receive neonatal resuscitation at birth

Inclusion Criteria:

* Inborn (not transferred to the hospital after birth)
* ≥34 weeks' gestation at birth, based on best obstetrical estimate
* Received PPV during neonatal resuscitation (as per provider's clinical assessment)

Exclusion Criteria:

* Congenital diaphragmatic hernia
* Airway anomalies

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36503 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Penetration of early SA rescue | Up to 2 years
  Proportion of eligible patients treated with SA as an early rescue device. Excludes SA after intubation attempt.

SECONDARY OUTCOMES:
Initial adoption of early SA rescue | Up to 2 years
  Quarters required to reach 10% penetration of SA use among eligible patients at hospital level
Sustainment of early SA rescue | Up to 1 year
  Proportion of SA use among eligible patients per quarter examined using linear mixed effects model to quantitatively assess successful sustainment (slope of penetration proportion positive or not significantly different than 0) versus decay (slope of penetration negative) post-implementation.

OTHER OUTCOMES:
Neonatal Intensive Care Unit (NICU) Admission | Up to 30 days of life
  Proportion of any admission to Neonatal Intensive Care Unit (NICU) before hospital discharge at hospital level, assessed among patients ≥35 weeks' Gestational Age (GA)
Hypoxic Ischemic Encephalopathy (HIE) | Up to 30 days of life
  Proportion of moderate to severe HIE at hospital level, assessed among patients ≥35 weeks' Gestational Age (GA)
Any exposure to Endotracheal Tube | Up to 30 days of life
  Proportion of any exposure to ventilation through Endotracheal Tube (ETT) prior to hospital discharge, including during resuscitation, at hospital level
Hospital Mortality | Up to 6 months of life
  Proportion of death before hospital discharge, at hospital level
Hospital length of stay | Up to 6 months of life
  Average days between birth and final disposition (death, transfer, or discharge), at hospital level

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Foglia, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (30):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rady Children's NICU at Rancho Springs Medical Center, Murrieta, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Jacobs Medical Center at University of California San Diego Health, San Diego, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - ChristianaCare, Newark, Delaware
  - St. John's Children's Hospital, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - MaineHealth Mid Coast Hospital, Brunswick, Maine
  - MaineHealth Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - South Shore University Hospital, Bay Shore, New York
  - Lenox Hill Hospital, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma Children's Hospital, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Parkland Health, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No